CLINICAL TRIAL: NCT07127653
Title: A 4-Week Lifting and Firming Efficacy Study Comparing a Retinol-Based Day Cream and a Lotion and Toner Bundle
Brief Title: Lotion and Toner Bundle 4-Week Lifting Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C25005018
Record Dates: First submitted 2025-08-01; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Lifting Efficacy; Facial Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retinol Day Cream Group (Experimental): Participants in this arm applied a retinol-based anti-wrinkle day cream to the full face for 4 weeks following a 3-week washout period. Assessments were conducted at baseline (T0), immediate post-use (Timm), and after 4 weeks of use (T4w). Evaluations included dermatologist lifting grade, DEEP imaging, and self-assessment questionnaire.
  Interventions: Other: Lotion and Toner Bundle
- Lotion and Toner Group (Experimental): Participants in this arm applied a lotion and toner bundle to the full face for 4 weeks following a 3-week washout period. Assessments were conducted at baseline (T0), immediate post-use (Timm), and after 4 weeks of use (T4w). Evaluations included dermatologist lifting grade, DEEP imaging, and self-assessment questionnaire.
  Interventions: Other: Retinol-Based Day Cream

INTERVENTIONS:
Other: Retinol-Based Day Cream — A commercially available day cream containing retinol and moisturizing ingredients. Applied twice daily (morning and evening) to the full face for 4 weeks.
  Arms: Lotion and Toner Group
Other: Lotion and Toner Bundle — A skincare regimen including a dermalift toner and a milky lotion. Applied twice daily (morning and evening) to the full face for 4 weeks.
  Arms: Retinol Day Cream Group

SUMMARY:
This is a single-center, parallel-arm, 4-week interventional study designed to evaluate the lifting and firming efficacy of two facial care regimens in middle-aged Chinese women. Participants were randomly assigned to use either a retinol-based day cream or a lotion-and-toner bundle. The study included dermatologist assessment, standardized facial photography, and self-assessment questionnaires. A total of 132 healthy women aged 45-55 with facial skin sagging were enrolled. The primary objective was to compare improvement in lifting grades after 4 weeks of product use. The trial was conducted at China-Norm Quality Technical Service Co., Ltd., in Shanghai, China.

DETAILED DESCRIPTION:
This 4-week study evaluated the efficacy of two skincare regimens on facial lifting and firmness in middle-aged Chinese women. Participants were randomly assigned to one of two arms: (1) retinol-based day cream or (2) a bundle of toner and lotion. The study included a 3-week wash-out period, followed by a 4-week treatment phase with full-face application. Assessments were conducted at T0 (baseline), Timm (immediate post-use), and T4w (end of 4-week use), using dermatologist grading (0-9 scale), DEEP imaging system, and self-reported questionnaires. Participants were required to avoid other skincare products during the study. A total of 132 subjects were enrolled; at least 80 completed clinical evaluation. The primary outcome was improvement in lifting grade from T0 to T4w; secondary outcomes included imaging analysis and subjective satisfaction. The study followed GCP principles and received ethical approval from the Ethics Committee at China-Norm. No serious adverse events were reported.

ELIGIBILITY:
Inclusion Criteria:

* 1. Chinese female with 45-55 years old. 2. All skin types (dry, normal, oily or mixed). 3. Regular users for toner, lotion and cream. 4. Self-claim with lack of firmness and has sagging concern. 5. Presenting with corresponding severity for the attribute evaluated by Dermatologist included:

  * Lifting (global face): 3≤grade≤6 (0-9 scale) 6. The BMI range should ≤24.9, and the BMI (BMI =Weight (kg)/ Height²(m²)) should remain stable within the range throughout the entire testing period. 7. Did not participate any clinical test or cosmetic product test on skin within 3 months.

    8. Did not participate any chemical procedures for previous 6 months and during the whole study.

    9. No disagreement of dermatologist because of other reasons that exclude the participation of the subject.

    10. In general, good health at the time of the study. 11. Willing and able to participate as evidenced by signing of informed consent & photo release form.

    12. Must be willing to comply with all study protocol requirements (pay attention: only use the skin care products provided during the study, not take topical or oral treatment like retinol, hormone, antioxidant health-care products which may affect the test product).

Exclusion Criteria:

* 1. Pregnant or breast-feeding woman or woman planning pregnancy during the study.

  2. Subject deprived of rights by a court or administrative order. 3. Major subject to a guardianship order. 4. Subject residing in a health or social care establishment. 5. Patient in an emergency setting. 6. Subject with a skin disease in the test areas as well as skin allergy (particularly e.g., acne, rosacea, eczema). 7. Subject presenting a stable or progressive serious disease (per investigator's assessment).

  8. Immuno-compromised subject. 9. Subject with history of allergy to cosmetic or personal care products or ingredients.

  10. Subject presenting excessive exposure to sunlight or UV radiation (investigator's assessment).

  11. Subject with history of sunlight sensitivity or allergies. 12. Subjects regularly practicing aquatic or nautical sports. 13. Subjects regularly attending a sauna. 14. Subject with physical highly sensitive constitution. 15. Subject with cardiovascular or circulatory history. 16. Subject with a history of skin cancer or malignant melanoma. 17. Intake of antihistamines, antibiotics, corticosteroids, non-steroidal anti-inflammatories or immune suppressants in the last 6 months before study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical Assessment by Dermatologist | Baseline and Week 4
  Lifting grade (0-9 scale) will be evaluated by dermatologist at T-3w, T0 (baseline), Timm and T4w.Six areas will be evaluated separately: eyebrow, upper eyelid, nasolabial zone, apple cheek, corner of mouth and jaw.

SECONDARY OUTCOMES:
Change in Facial Wrinkle Depth Measured by Standardized Digital Photography and Image Analysis Software | Baseline and Week 4
Questionnaire | Baseline and Week 4
  Change in self-reported score for skin smoothness and softness from baseline to week 4, based on 5-point Likert scale questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai 200072, Shanghai, China

IPD SHARING:
Plan to Share IPD: No